CLINICAL TRIAL: NCT00692497
Title: Costs-effectiveness and Waiting Time for Direct Electronic Referral and Booking of Outpatient Day Case Surgery Compared With Traditional Referral Routines. A Randomised Controlled Trial
Brief Title: Electronic Referral and Booking of Outpatient Day Case Surgery Compared With Traditional Referral Routines.
Acronym: one-stop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: P REK NORD 122/2006
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Referral and Consultation; Telemedicine; Surgery, Outpatient; Surgery, Day; Medical Records Systems, Computerized; Health Services Research; Health Care Surveys
Keywords: One-Stop; Public Health Research; Delivery of Health Care/*standards; Evaluation Studies; Referral; Surgery, Outpatient; Surgery, Day; Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): The one stop strategy is a set of interventions directed at GPs referring to the University Hospital. The interventions include: Guidelines for referral, standardised electronic referrals, booking for outpatient surgery and a patient information form.
  Interventions: Behavioral: one stop (Electronic standardised referrals and appointment bookings)
- 2 (No Intervention): Patients in the control group are randomised to use the regular patient pathway prior to day case outpatient surgery. All these patients are referred to the surgical outpatient clinic. At the outpatient clinic patients are examined by a surgeon and indications for surgery is decided by the surgeon. If indicated, patients are then referred to outpatient surgery and the surgical procedure is performed several weeks after the examination.

INTERVENTIONS:
Behavioral: one stop (Electronic standardised referrals and appointment bookings) — The one stop strategy is a set of interventions directed at GPs referring to the University Hospital. The interventions include: Guidelines for referral, standardised electronic referrals, booking for outpatient surgery and a patient information form.
  Arms: 1

SUMMARY:
We want in this study to investigate the cost-effectiveness and waiting time of direct electronic referral and booking of outpatient surgery compared to the traditional patient pathway where the patient is seen at the outpatient clinic prior to surgery.

DETAILED DESCRIPTION:
Waiting time from referral to day case outpatient surgery is unacceptable long. In Norway it is as much as 48 weeks for common conditions like gallstones, inguinal hernia and sinus pilonidalis. Electronic standardised referrals sent by the Norwegian Healthcare Network, and booking of surgery by the general practitioner might be a way to reduce the waiting time and increase the cost effectiveness of outpatient surgery.

The trial is designated as a randomized controlled trial were selected patients (inguinal hernia, gall stone disease and sinus pilonoidalis) referred to the university hospital, were either randomized to direct electronic referral and booking for outpatient surgery (one stop), or using the traditional patient pathway where all patients are seen at the outpatient clinic several weeks before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible if they were diagnosed by their GP for an inguinal hernia, sinus pilonidalis or gallstone disease which require surgical treatment.

Exclusion Criteria:

* Patients with medical conditions making them unfit for outpatient surgery admitted to the surgical department prior to surgery are not eligible

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-10; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
waiting time | one year

SECONDARY OUTCOMES:
cost effectiveness | one year

CONTACTS AND LOCATIONS:
Overall Officials: Rolv-Ole Lindsetmo, MD, PhD, Principal Investigator — University of Tromso; Roar Johnsen, MD, PhD, Prof., Study Chair — University of North Norway; Knut M Augestad, MD, Study Director — Norwegian Centre for Telemedicine and Department of Gastrointestinal Surgery, University Hospital of North Norway, Norway
Locations (1):
- Norwegian Centre of Telemedicine, Tromsø, Norway

REFERENCES:
- [Derived] Augestad KM, Revhaug A, Vonen B, Johnsen R, Lindsetmo RO. The one-stop trial: does electronic referral and booking by the general practitioner (GPs) to outpatient day case surgery reduce waiting time and costs? A randomized controlled trial protocol. BMC Surg. 2008 Aug 11;8:14. doi: 10.1186/1471-2482-8-14. PMID 18694477